CLINICAL TRIAL: NCT03026478
Title: A Comparative Study on Clinical Efficacy of Clobetasol and Betamethasone in Orabase in Combination With Clotrimazole, in Oral Lichen Planus
Brief Title: Topical Betamethasone and Clobetasol in Orabase in Oral Lichen Planus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Garlapati Komali (Other)
Responsible Party: Sponsor-Investigator, Garlapati Komali, PROFESSOR, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Organization: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMVIDS&RC/IEC/OMR/DN/0003-15
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; betamethasone; clobetasol; orabase
MeSH Terms: conditions — Lichen Planus, Oral | interventions — betamethasone-17,21-dipropionate; Gels; Clobetasol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betamethasone dipropionate 0.05% (Experimental): topical Betamethasone dipropionate 0.05% in orabase with clotrimazole 1% in oral lichen planus two times a day for one month
  Interventions: Drug: Betamethasone Dipropionate
- Clobetasol propionate 0.05% (Active Comparator): Topical Clobetasol propionate 0.05% in orabase with clotrimazole 1% in oral lichen planus patients two times a day for a month
  Interventions: Drug: Clobetasol Propionate

INTERVENTIONS:
Drug: Betamethasone Dipropionate
  Other Names: Betamethasone Dipropionate 0.05% gel
  Arms: Betamethasone dipropionate 0.05%
Drug: Clobetasol Propionate
  Other Names: Clobetasole Propionate 0.05% gel
  Arms: Clobetasol propionate 0.05%

SUMMARY:
Oral Lichen Planus (OLP) is an autoimmune, chronic inflammatory mucocutaneous disease characterized by pain and burning sensation. The major types of OLP are the following: reticular, atrophic, erosive-ulcerative, bullous and pigmentous form.Its etiology remains unclear. The presence of auto-cytotoxic T cell clones in the lesions suggests the role of autoimmunity. Numerous treatment options of OLP include topical and systemic agents depending on severity of lesions . Topical corticosteroids abide the mainstay of therapy,and are widely accepted as the primary treatment of choice.Hence this study is designed to evaluate and compare the clinical efficacy of topical Clobetasol 0.05% in orabase and Betamethasone 0.05% in orabase in combination with Clotrimazole 1% in the management of symptomatic Oral Lichen Planus.

DETAILED DESCRIPTION:
Patients of either sex, irrespective of age attending the Department of Oral Medicine & Radiology, Panineeya Mahavidhyalaya Institute of Dental Sciences and Research Centre, Hyderabad who are clinically and histopathologically diagnosed with Oral Lichen Planus shall be included in the study group after obtaining an informed consent from the patients.

Study design: Prospective study.

Sample size:

A total of 30 patients will be randomly divided into 2 groups with 15 patients in each group.

Methodology:

30 patients who are diagnosed with Oral Lichen Planus by clinical and histopathological examination will be randomly assigned into 2 drug groups and burning sensation will be assessed by VAS Scale and also clinical improvement will be assessed at interval of 1 week till 4 weeks.

GROUP A: This group of patients will receive topical Clobetasol 0.05% in orabase and Clotrimazole 1%.

GROUP B: This group of patients will receive topical Betamethasone 0.05% in orabase and Clotrimazole 1%.

Inclusion criteria:

1. Patients with Oral Lichen Planus, who are willing to participate in the study.
2. Patients who are physically healthy and well oriented in time, space and as a person.
3. Patients clinically and histopathologically diagnosed with Oral Lichen Planus.
4. Patients with symptoms i.e. pain and burning sensation due to oral lichen planus.

Exclusion Criteria :

1. Patients with Oral Lichen Planus, who are not willing to participate in the study.
2. Patients with any other mucosal disease or any other skin disease which may be associated with oral lesions.
3. Patients with a known allergy or contraindication to study medications.
4. Patients with systemic diseases, where steroids are contraindicated.
5. Pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Oral Lichen Planus, who are willing to participate in the study.
2. Patients who are physically healthy and well oriented in time, space and as a person.
3. Patients clinically and histopathologically diagnosed with Oral Lichen Planus.
4. Patients with symptoms i.e. pain and burning sensation due to oral lichen planus.

Exclusion Criteria:

1. Patients with Oral Lichen Planus, who are not willing to participate in the study.
2. Patients with any other mucosal disease or any other skin disease which may be associated with oral lesions.
3. Patients with a known allergy or contraindication to study medications.
4. Patients with known history of systemic diseases, where steroids are contraindicated.
5. Pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05-06 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Based on Visual analog scale and size of the lesion | Each patient will be assessed for a total time frame of 1 month at a regular interval of 1 week.
  study is in progress

CONTACTS AND LOCATIONS:
Overall Officials: KOMALI GARLAPATI, Principal Investigator — PMVIDS & RC
Locations (1):
- Komali Garlapati, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No